CLINICAL TRIAL: NCT02870556
Title: Effect of Cervical Epidural Analgesia on the Occurrence of Pharyngocutaneous Fistula Following Salvage Laryngectomy and Reconstruction With Pectoralis Major Myocutaneous Flap
Brief Title: Effect of Cervical Epidural Analgesia on the Occurrence of Pharyngocutaneous Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Not yet assigned
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Cutaneous Fistula; Laryngectomy
Keywords: cervical epidural, laryngectomy, pharyngocutaneous fistula
MeSH Terms: conditions — Cutaneous Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EP, Cervical epidural group (Experimental): patients undergoing salvage laryngectomy (failed radiotherapy to treat laryngeal cancer) will receive cervical epidural analgesia in addition to the standard general anesthesia (induction with propofol 2 mg / kg, endotracheal intubation facilitated by cis-atracurium 0.3 mg / kg and 0.15 mg /kg on demand and maintained with inhalational anesthetic sevoflurane) Cervical epidural technique: epidural needle will be inserted at C 6-C7 or C7-T1 under fluoroscopy in prone position, 6 ml of 0.125% bupivacaine and fentanyl 2 mic/ ml will be administered before skin incision followed by 4 ml of the same injectate, will be infused continously for 2 days
  Interventions: Device: cervical epidural analgesia
- GA, General anesthesia (Active Comparator): patients undergoing salvage laryngectomy (failed radiotherapy to treat laryngeal cancer) will receive standard general anesthesia only (induction with propofol 2 mg / kg, endotracheal intubation facilitated by cis-atracurium 0.3 mg / kg and 0.15 mg /kg on demand and maintained with inhalational anesthetic sevoflurane) in addition to postoperative analgesia through patient controlled intravenous morphine analgesia (PCA), that involve 1 mg continuous infusion and 2 mg boluses with lockout interval 10 min
  Interventions: Device: cervical epidural analgesia

INTERVENTIONS:
Device: cervical epidural analgesia

SUMMARY:
Pharyngocutaneous fistula (PCF) is the most commonly reported postoperative complication in total laryngectomy patients. PCF significantly increases morbidity, length of hospitalization, and cost of care, in addition to delaying the beginning of adjuvant therapy. The reported incidence of PCF ranges from 3% to 65%.The increased use of radiation in the primary management of laryngeal carcinoma has resulted in an increase in the PCF formation after salvage laryngectomy (STL).

Previously reported risk factors for PCF development include preoperative radiotherapy, tumor stage, concomitant neck dissection, prior need for tracheotomy, hypoalbuminemia and anemia.

Among surgical options, the pectoralis major myofascial flap has been proposed to cover the pharyngeal closure, to interpose non-irradiated tissue between the neopharynx and the skin during STL. Nonetheless, the efficacy of this approach is not fully established.Epidural anesthesia improves the blood supply due to its vasodilating effect. The aim of the study is to evaluate the effect of perioperative cervical epidural analgesia on the occurrence of pharyngocutaneous fistula following salvage laryngectomy and reconstruction with pectoralis major myocutaneous flap.

DETAILED DESCRIPTION:
Patients will be divided into two equal groups, group (EP), will receive perioperative cervical epidural analgesia in addition to general anesthesia and group (GA) will receive general anesthesia and postoperative analgesia through patient controlled intravenous morphine analgesia (PCA), that involve 1 mg continuous infusion and 2 mg boluses with lockout interval 10 min.

Cervical epidural technique: epidural needle will be inserted at C 6-C7 or C7-T1 under fluoroscopy in prone position, 6 ml of 0.125% bupivacaine and fentanyl 2 mic/ ml will be administered before skin incision followed by 4 ml of the same injectate, will be infused continously for 2 days

ELIGIBILITY:
Inclusion Criteria:

* Patients who failed treatment with radiotherapy for laryngeal cancer

Exclusion Criteria:

1. Infection at the site of flap
2. Primary laryngectomy without radiotheraapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2016-12-20 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
pharyngocutaneous fistula following salvage laryngectomy and reconstruction with pectoralis major myocutaneous flap | 2 weeks postoperatively

SECONDARY OUTCOMES:
Pain intensity measured by visual analogue scale (VAS) | 0 h (immediately postoperative), 2h, 6h, 12h, 24h, 48h (postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Diab, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided